CLINICAL TRIAL: NCT04459715
Title: A Randomized, Double-Blind Placebo-Controlled, Phase 3 Study of Debio 1143 in Combination With Platinum-Based Chemotherapy and Standard Fractionation Intensity-Modulated Radiotherapy in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck, Suitable for Definitive Chemoradiotherapy (TrilynX)
Brief Title: A Study of Xevinapant (Debio 1143) in Combination With Platinum-Based Chemotherapy and Standard Fractionation Intensity-Modulated Radiotherapy in Participants With Locally Advanced Squamous Cell Carcinoma of the Head and Neck, Suitable for Definitive Chemoradiotherapy (TrilynX)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has crossed the pre-defined futility boundary at the Interim Analysis.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: GORTEC (Head and Neck Oncology and Radiotherapy Group) (Unknown); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS202359_0006; 2020-000377-25 (EudraCT Number); Debio 1143-SCCHN-301 (Other: Previous Sponsor Identifier)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: TrilynX
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xevinapant (Debio 1143) (Experimental): Participants received:
  Concomitant chemo-radiation therapy period (Cycles 1-3):
  * Radiotherapy
  * Cisplatin
  * Xevinapant (Debio 1143)
  Monotherapy period (Cycles 4-6):
  • Xevinapant (Debio 1143)
  Interventions: Drug: Xevinapant (Debio 1143); Drug: Cisplatin; Radiation: Intensity Modulation Radiation Therapy (IMRT)
- Placebo (Active Comparator): Participants received:
  Concomitant chemo-radiation therapy period (Cycles 1-3):
  * Radiotherapy
  * Cisplatin
  * Matched placebo
  Monotherapy period (Cycles 4-6):
  • Matched placebo
  Interventions: Drug: Cisplatin; Radiation: Intensity Modulation Radiation Therapy (IMRT); Drug: Placebo

INTERVENTIONS:
Drug: Xevinapant (Debio 1143) — Xevinapant (Debio 1143) administrated as oral solution from Day 1 to 14, every 21-day cycle.
  Arms: Xevinapant (Debio 1143)
Drug: Cisplatin — Cisplatin administered as an IV infusion every 3 weeks (Q3W).
Radiation: Intensity Modulation Radiation Therapy (IMRT) — 70 Gy given in 35 fractions over 7 weeks.
Drug: Placebo — Matched placebo administrated as oral solution from Day 1 to 14, every 21-day cycle.
  Arms: Placebo

SUMMARY:
The primary objective of the study was to demonstrate superior efficacy of Xevinapant (Debio 1143) vs placebo when added to chemoradiotherapy (CRT) in locally advanced squamous cell carcinoma of the head and neck (LA-SCCHN).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1
* Histologically confirmed diagnosis of previously untreated Locally Advanced Squamous Cell Carcinoma of the Head and Neck (LA-SCCHN) participant (stage III, IVa or IVb according to the American Joint Committee on Cancer(AJCC))/Classification of malignant tumors: T=size of the primary tumor, N=regional lymph node involvement, M=distant metastasis (TNM) Staging System, 8th Edition.) suitable for definitive ChemoRadiotherapy (CRT), of at least one of the following sites: oropharynx, hypopharynx and larynx
* For OroPharyngeal Cancer (OPC) participants, primary tumors must be human papillomavirus (HPV)-negative as determined by p16 expression using immunohistochemistry
* Evaluable tumor burden (measurable and/or non-measurable tumor lesions) assessed by computed tomography scan (CT-scan) or magnetic resonance imaging (MRI), based on Response evaluation criteria in solid tumors (RECIST) version 1.1
* Peripheral neuropathy less than (<) grade 2
* Adequate hematologic, renal and hepatic function
* Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* Primary tumor of nasopharynx, paranasal sinuses, nasal or oral cavity, salivary, thyroid or parathyroid gland pathologies, skin or unknown primary site
* Metastatic disease (stage IVc as per AJCC/TNM, 8th Ed.)
* Prior definitive or adjuvant Radiotherapy (RT) and/or radical surgery to the head and neck region which may jeopardize the primary tumor irradiation plan, or any other prior SCCHN systemic treatment, including investigational agents
* Documented weight loss of >10% during the last 4 weeks prior to randomization (unless adequate measures are undertaken for nutritional support), OR plasmatic albumin < 3.0 g/dL. No albumin transfusions are allowed within 2 weeks before randomization
* Known allergy to Xevinapant (Debio 1143), cisplatin, carboplatin, other platinum-based agent or any excipient known to be present in any of these products or in the placebo formulation
* other protocol defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (288):
- United States (44):
  - The University of Alabama at Birmingham - Hazelrig-Salter Radiation Oncology Center (HSROC), Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Regents of the University of California, San Francisco, California
  - UCSF, San Francisco, California
  - The Oncology Institute of Hope & Innovation, Whittier, California
  - University of Colorado at Denver and Health Sciences Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Lombardi Comprehensive Cancer Center, Georgetown University Medical Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - ASCLEPES Research Centers, Weeki Wachee, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - IACT Health, John B. Amos Cancer Center, Columbus, Georgia
  - Inventa Center for Cancer Research At Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky, Brownsboro Hospital Campus, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess (BI Lahey)/Harvard Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University South Hospital, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Karmanos Cancer institute, Detroit, Michigan
  - University of Missouri - Ellis Fischel Cancer Center, Columbia, Missouri
  - MidAmerica Cancer Care, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Center of Nevada (Southern Hills) (USA), Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NYU Langone Hospital-Long Island Oncology, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYU Grossman School of Medicine, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center- Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina- Hollings Cancer Center, Charleston, South Carolina
  - MD Anderson, Houston, Texas
  - IHO Corporation/Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
- Argentina (5):
  - Hospital Aleman, Buenos Aires
  - Instituto Medico Especialazado Alexander Fleming, Buenos Aires
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Instituto de Oncologia de Rosario, Santa Fe
  - Clinica Viedma, Viedma
- Australia (6):
  - Ashford Cancer Centre Research, Tennyson Centre, Adelaide
  - St Vincents Hospital, Darlinghurst
  - St Vincents Hospital Melbourne, Fitzroy
  - Peter MacCallum Cancer Centre, Melbourne
  - Wollongong Hospital, Wollongong
  - Princess Alexandra Hospital, Cancer Trials Unit, Woolloongabba
- Austria (4):
  - Klinische Abteilung fur Allgemeine HNO Universitatsklinik fur Hals-, Nasen- und Ohrenheilkunde, Graz
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitätsklinik für Innere Medizin III der PMU, Salzburg
  - Medical University of Vienna, Department of Medicine I, Division of Oncology, Vienna
- Belgium (10):
  - Cliniques universitaires Saint-Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent UZ Gent, Ghent
  - Hopital de Jolimont, Rue Ferrer, La Louvière
  - UZ Leuven, Radiotherapy & Oncology, Leuven
  - Centre Hospitalier de l'Ardenne (CHA), Libramont
  - CHU UCL Namur Site Sainte Elisabeth, Namur
  - A.Z. Nikolaas, Sint-Niklaas
  - GZA Sint-Augustinus, Wilrijk
- Brazil (11):
  - Fundação Pio XII- Hospital de Cancer de Barretos, Rua Antenor Duarte Vilela, Barretos
  - Hospital de Caridade de Ijui, Avenida David Jose Martins, Ijuí
  - Liga Norte Riograndense Contra o Câncer, Avenida Miguel Castro, Natal
  - Centro Gaúcho Integrado, Rua Costa, Porto Alegre
  - Hospital Santa Rita Centro de Pesquisa Clínica Novos Tratamentos Em Câncer, Porto Alegre
  - Hospital Santa Rita, Centro de Pesquisa Clínica Novos Tratamentos Em Câncer, Porto Alegre
  - National Cancer Institute, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia - FMABC - Faculdade de Medicina do ABC, Santo André
  - Hospital de Base de Sao Jose do Rio Preto, Av. Brigadeiro Faria Lima, São José do Rio Preto
  - Instituto do Cancer do Estado de Sao Paulo (ICESP), São Paulo
  - Oswaldo Cruz German Hospital, São Paulo
- Canada (6):
  - London Regional Cancer Program, London Health Sciences Centre, London
  - CHU Montréal, Montreal
  - CIUSSS de l'Est de l'Ile de Montreal - Hopital Maisonneuve-Rosemont, Montreal
  - Hopital Maisonneuve-Rosemont, Montreal
  - CHU de Quebec-Université Laval, Québec
  - Sunnybrook Research Institute, Toronto
- China (21):
  - Beijing Cancer Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - The 5th Affiliated Hospital of Sun yet-sen university, Guangdong
  - The 2nd Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Province Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning
  - Lin Yi Cancer Hospital, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai
  - Shantou University Cancer Hospital, Shantou
  - Liaoning Cancer Hospital & institute, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tongji Hospital/Tongji Medical College, Huazhong University of Science, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- Czechia (4):
  - University Hospital hradec Kralové, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava-Poruba
  - Hospital Na Bulovce, Prague
  - KOC KNTB a.s. Zlín, Zlín
- France (30):
  - CHU Amiens Picardie - Hopital Sud, Amiens
  - Institut de Cancérologie de l Ouest (ICO), Angers
  - Institut Sainte Catherine, Avignon
  - Centre hospitalier Universitaire de Bordeaux, Bordeaux
  - CHRU de Brest Hopital Morvan, Brest
  - Centre Jean Perrin CLCC, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Centre Guillaume Le Conquerant, Le Havre
  - Clinique Victor Hugo, Le Mans
  - Centre hospitalier Libourne, Libourne
  - Centre Oscar Lambret, Lille
  - Hôpital du Scorff, Lorient
  - Centre Leon Berard, Lyon
  - Service d'Oncologie Médicale, CHU Timone, Marseille
  - Hôpital Nord Franche Comté, Montbéliard
  - Institut Regional du Cancer de Montpellier, Montpellier
  - LHopital prive du Confluent Nantes, Nantes
  - CCConcorde (GCS), Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - CHU Nimes, Nîmes
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel CLCC, Rouen
  - CHP Saint Gregoire FINESS, Saint-Grégoire
  - Institut de Cancérologie de l'Ouest - Site Saint Herblain, Saint-Herblain
  - ICANS, Strasbourg
  - Institut Claudius Regaud - IUCT-O, Toulouse
  - CHU de Tours, Tours
  - The Public Hospital L'Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy - Service de radiotherapie, Villejuif
- Georgia (8):
  - Evex Hospitals Oncology Center, Kutaisi
  - Academician Fridon Todua Medical Center-Ltd Research Institute of Clinical Medicine, Tbilisi
  - Cancer Research Cent 4, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - JSC "Evex Hospitals", Tbilisi
  - LEPL First University Clinic of Tbilisi State Medical University, Tbilisi
  - New Hospitals, Tbilisi
  - Simon Khechinashvili University Clinic, Tbilisi
- Germany (12):
  - CAMPUS CHARITÉ MITTE, Klinik f.Strahlentherapie, Berlin
  - Charité - Universitätsmedizin Berlin Campus Virchow, Berlin
  - Strahlenklinik des Uni-Klinikums, Erlangen
  - Department of radiation oncology, University Hospital Essen, Essen
  - Univesitätsklinikum Essen (AöR) Klinikum und Poliklinik für Strahlentherapie, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Jena - Klinik fuer Hals - Nasen und Ohrenheilkunde HNO, Jena
  - University Medical Center Schleswig-Holstein, Campus Kiel, Kiel
  - Universitatsklinikum Leipzig AoR, Klinik für Strahlentherapie, Leipzig
  - Universitaetsmedizin Mannheim UMM, Klinik fuer Hals-Nasen-Ohrenheilkunde Kopf- und Halschirurgie, Mannheim
  - Universitaetsklinikum Regensburg, Regensburg
  - Universitaetsmedizin Rostock, Rostock
- Greece (3):
  - Agioi Anargiroi General Oncology Hospital of Kifissia, Athens
  - Attikon University Hospital, Athens
  - Theagenio Anticancer Hospital, Thessaloniki
- Hungary (5):
  - Orszagos Onkologiai Intezet Sugarterapias Osztaly, Budapest
  - Uzsoki Utcai Korhaz Onkologiai Osztaly, Budapest
  - Petz Aladár Megyei Kórház Onkoradiológiai Osztály, Győr
  - Pecsi Tudomanyegyetem Klinikai Kozpont Onkoterapias Intazet, Pécs
  - Szegedi Tudományegyetem ÁOK Onkoterápiás Klinika, Szeged
- Israel (4):
  - Rambam Healthcare Campus, Haifa
  - Research Fund of the Hadassah Medical Organization, Jerusalem
  - Rabin Medical Center, Petach Tiqva
  - Sheba Medical Center, Ramat Gan
- Italy (19):
  - Centro di Riferimento Oncologico, Aviano
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia, Brescia
  - Istituto di Candiolo IRCCS, Candiolo
  - Azienda Sanitaria Ospedaliera Santa Croce e Carle - Oncologia Medica -Ospedale Carle, Cuneo
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - IRCCS AOU San Martino, Genova
  - Ospedale "Vito Fazzi" Lecce, Lecce
  - Az. USL 6 Ospedali Riuniti-Ospedale di Livorno, Livorno
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola
  - IRCCS-Istituto Europeodi Oncologia The European Institute of Oncology IEO, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Policlinico di Modena, Modena
  - AORN Ospedale dei Monaldi, Napoli
  - AOU "Luigi Vanvitelli", Napoli
  - Istituto Nazionale Tumori (INT) IRCCS Fondazione "G. Pascale", Napoli
  - Istituto Oncologico Veneto Irccs, Padua
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome
  - ASL2_Presidio Ospedaliero San Paolo, Savona
- Japan (14):
  - National Cancer Center Hospital East, Chiba
  - National Cancer Center Hospital, Chuo-ku Tokyo
  - Saitama Medical University International Medical Center, Hidaka
  - Hyogo Cancer Center, Hyōgo
  - University Hospital Kyoto Prefectural University of Medicine, Kamigyō-ku
  - Tokai University Hospital, Kanagawa
  - Hokkaido University Hospital, Kita-ku
  - Okayama University Hospital, Kita-ku
  - Kobe University Hospital, Kobe
  - Cancer Institute Hospital of JFCR, Kōtoku
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Shizuoka Cancer Center, Nagaizumi-cho
  - Osaka International Cancer Institute, Osaka
  - Tokyo Medical University Hospital, Tokyo
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne - Klinika Onkologii i Radioterapii, Gdansk
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Centrum Onkologii- Instytut im. Marii Sklodowskiej-Curie Oddzial w Gliwicach, Gliwice
  - NZOZ Provita Prolife Centrum Medyczne, Lodz
  - SP ZOZ MSWiA z W-M CO w Olsztynie, Olsztyn
- Portugal (9):
  - Centro Clinico Academico, Braga
  - Hospital de Braga, Braga
  - Instituto Português de Oncologia de Coimbra Francisco Gentil, EPE, Coimbra
  - Centro Hospitalar Universitário do Algarve - Hospital de Faro (PRT), Faro
  - Centro Hospitalar Universitário Lisboa Norte, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, Porto
  - Centro Hospitalar Universitario São João, Porto
  - Hospital Pedro Hispano, Porto
  - Instituto Portugues de Oncologia Porto Francisco Gentil, E.P.E, Porto
- Russia (10):
  - State Autonomous Healthcare Institution "Republican Clinical Oncological Dispensary of the Ministry of Healthcare of the Republic of Tatarstan", Kazan'
  - Krasnoyarsk Regional Clinical Oncological Dispensary named after A.I.Kryzhanovsky, Krasnoyarsk
  - Kursk Regional Clinical Oncology Dispensary, Kursk
  - FGBU N.N.Blokhin Russian Cancer Research Center, Moscow
  - EuroCityClinic, Saint Petersburg
  - FSBI National Med Research Cancer Center N.N. Petrov, Saint Petersburg
  - Saint- Petersburg Clinical Research Center of Specialized Types of Medical Care (Oncology), Saint Petersburg
  - Republican Clinical Oncological Dispensary of Bashkortostan, Ufa
  - State Budgetary Healthcare Institution Republican Clinical Oncology Dispensary (RUS), Ufa
  - State Budgetary Institution of Healthcare of Yaroslavl region Clinical oncology hospital, Yaroslavl
- South Korea (9):
  - Pusan National University Hospital, Busan
  - National Cancer Center Hematologic Oncology, Goyang-si
  - National Cancer Center, Goyang-si
  - Asan Medical Center, Asian Cacer Center, Seoul
  - Asan Medical Center, Seoul
  - KonKuk University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Oncol & Hematology, Yangsan
- Spain (25):
  - Fundacion Centro Oncologico de Galicia (COG) "Jose Antonio Quiroga y Pineyro", A Coruña, Galicia
  - Fundacin Oncolgico de Galicia Jos Antonio Quiroga y Pieyro, A Coruña
  - Hospital Clinic Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia Badalona, Barcelona
  - Institut Català d'Oncologia, Hospital Duran, Barcelona
  - Institut Universitari Dexeus-Quiron (ESP), Barcelona
  - Hospital Reina Sofía, Córdoba
  - Institut Català d'Oncologia, Girona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Clinica Universidad de Navarra, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario La Paz, Madrid
  - Althaia, Xarxa Assistencial, Manresa
  - Fundacio Althaia, Manresa
  - Hospital Civil (Hospital Regional Universitario), Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Marqués de Valdecilla. Santander, Santander
  - Fundacion Investigacion Hospital General Universitario de Valencia FiHgU (ESP), Valencia
  - Hospital Universitario La Fe, Valencia
  - IVO, Valencia
- Switzerland (3):
  - Inselspital, Bern University Hospital, Universitätsklinik für Radio-Onkologie, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne
- Taiwan (7):
  - Chang-Gung Memorial Hospital-Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital (VGHTP), Taipei
  - Chang Gung Medical Foundatoin Linkou Chang Gung Memorial Hospital, Taoyuan
- Ukraine (3):
  - Medical center ASKLEPION LLC, Khodosovka
  - Kiev City Clinical Oncology Centre, Kiev
  - Medical center of Yuriy Spizhenko, Soborna Vulytsia, Kyiv
- United Kingdom (11):
  - Aberdeen Royal infirmary, Dept. of Oncology, Aberdeen
  - Royal Marsden NHS Foundation Trust, Chelsea
  - NHS Greater Glasgow and Clyde, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Mount Vernon Cancer Centre, Northwood
  - Nottingham University Hospitals NHS Trust, Nottingham
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - The Royal Marsden NHS Foundation Trust - Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
URL: http://bit.ly/IPD21

REFERENCES:
- [Derived] Bourhis J, Licitra LF, Burtness B, Psyrri A, Haddad R, Harrington K, Cohen EEW, Tao Y, Tiscoski KA, Matitashvili A, Tahara M, Sukari A, Rutkowski T, Salas S, Nauwelaerts H, Scheerlinck R, Ha NT, Schroeder A, Rodriguez-Gutierrez A, Schoenfeld JD. Xevinapant or Placebo Plus Platinum-Based Chemoradiotherapy in Unresected Locally Advanced Squamous Cell Carcinoma of the Head and Neck (TrilynX): A Randomized, Phase III Study. J Clin Oncol. 2025 Oct 10;43(29):3209-3220. doi: 10.1200/JCO-25-00272. Epub 2025 Sep 3. PMID 40902136
- [Derived] Bourhis J, Burtness B, Licitra LF, Nutting C, Schoenfeld JD, Omar M, Bouisset F, Nauwelaerts H, Urfer Y, Zanna C, Cohen EE. Xevinapant or placebo plus chemoradiotherapy in locally advanced squamous cell carcinoma of the head and neck: TrilynX phase III study design. Future Oncol. 2022 May;18(14):1669-1678. doi: 10.2217/fon-2021-1634. Epub 2022 Feb 17. PMID 35172587
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Debio 1143 + CRT: Participants received a combination of Debio 1143 along with Chemoradiotherapy (CRT): Radiotherapy +Cisplatin + Xevinapant (Debio 1143). Participants received 6 cycles of oral solution of Xevinapant at a dose of 200 milligrams per day (mg/day) once daily from Day 1 to 14, per 3-week cycle in combination with 70 Gray (Gy) of intensity modulated radiation therapy (IMRT) in 35 fractions, 2 Gy/fraction, over 7 weeks, and High-dose cisplatin (100 Milligram per square meter (mg/m2)) on Day 2 of a 3-week cycle per 3 cycles (combination therapy period). If high-dose cisplatin 100 mg/m2 was not tolerated after the first dose, participants could be switched to carboplatin (10 Milligrams per milliliter (mg/mL), intravenous (iv) infusion), followed by 3 cycles of monotherapy of Xevinapant at a dose of 200 mg/day from Day 1 to 14, per 3-week cycle (monotherapy period).
- Sequence 2: Placebo + CRT: Participants received a combination of placebo matched to Debio 1143 along with Chemoradiotherapy(CRT): Radiotherapy +Cisplatin+ placebo matched to Xevinapant (Debio 1143). Participants received 6 cycles of oral solution of placebo matched to Xevinapant once daily from Day 1 to 14, per 3-week cycle in combination with 70 Gray (Gy) of intensity modulated radiation therapy (IMRT) in 35 fractions, 2 Gy/fraction, over 7 weeks, and High-dose cisplatin (100 mg/m2) on Day 2 of a 3-week cycle per 3 cycles(combination therapy period).If high-dose cisplatin 100 mg/m2 was not tolerated after the first dose, participants could be switched to carboplatin (10mg/mL, iv infusion), followed by 3 cycles of monotherapy of placebo matched to Xevinapant from Day 1 to 14, per 3-week cycle (monotherapy period).
Period: Overall Study
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Started | 364 | 366
Completed | 0 | 0
Not Completed | 364 | 366
Not completed — Adverse Event | 3 | 3
Not completed — Death | 111 | 93
Not completed — Lost to Follow-up | 10 | 9
Not completed — Other Reasons | 4 | 5
Not completed — PROTOCOL DEVIATION | 0 | 1
Not completed — RANDOMIZED BY MISTAKE | 0 | 1
Not completed — STUDY TERMINATED BY SPONSOR | 214 | 232
Not completed — Withdrawal by Subject | 22 | 22

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Debio 1143 + CRT: Participants received a combination of Debio 1143 along with Chemoradiotherapy (CRT): Radiotherapy +Cisplatin + Xevinapant (Debio 1143). Participants received 6 cycles of oral solution of Xevinapant at a dose of 200 milligrams per day (mg/day) once daily from Day 1 to 14, per 3-week cycle in combination with 70 Gray (Gy) of intensity modulated radiation therapy (IMRT) in 35 fractions, 2 Gy/fraction, over 7 weeks, and High-dose cisplatin (100 mg/m2) on Day 2 of a 3-week cycle per 3 cycles (combination therapy period). If high-dose cisplatin 100 mg/m2 was not tolerated after the first dose, participants could be switched to carboplatin (10mg/mL, iv infusion), followed by 3 cycles of monotherapy of Xevinapant at a dose of 200 mg/day from Day 1 to 14, per 3-week cycle (monotherapy period).
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT | Total
Number analyzed (Participants) | 364 | 366 | 730
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (8.01) | 60 (8.53) | 60 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 57 | 121
  Male | 300 | 309 | 609
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Hispanic or Latino | 41 | 46 | 87
  Ethnicity-Not Hispanic or Latino | 264 | 273 | 537
  Ethnicity-Unknown or Not Reported | 59 | 47 | 106
  Race-Asian | 59 | 60 | 119
  Race-Black or African American | 5 | 6 | 11
  Race-Other | 5 | 9 | 14
  Race-Unknown or Not Reported | 42 | 35 | 77
  Race-White | 253 | 256 | 509

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to the date of death. Calculated via Kaplan Meier method.
Time Frame: From randomization to the earliest between death or EOS (up to 188 weeks and 5 days)
Population: The ITT set included all randomized participants. Participants were analyzed according to the randomized treatment (assigned arm) assignment following the intention-to-treat principle.
Measure: Median (Full Range); unit: months
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 366
months | NA [0.0 to 37.6] — Due to the limited number of events, the median could not be derived. | NA [0.0 to 39.4] — Due to the limited number of events, the median could not be derived.

2. Secondary Outcome: Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as Assessed by Blinded Independent Review Committee (BIRC)
Description: PFS according to RECIST v1.1 defined as the time from randomization to the first occurrence of progression (radiological or clinical, as assessed by the BIRC) or death from any cause. According to RECIST 1.1, progressive disease (PD) was defined as a 20% relative increase in the sum of diameters (SOD) of target lesions, taking as reference the nadir SOD and an absolute increase of >5 millimeter (mm) in the SOD, or the appearance of new lesions. Calculated via Kaplan Meier method.
Time Frame: From randomization to the first occurrence of progression (radiological or clinical, as assessed by the BIRC) or death from any cause or EOS (up to 188 weeks and 5 days )
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 366
months | 26.8 [15.93 to NA] — Due to the limited number of events, the upper limit of the 95% CI for the median could not be derived. | 33.1 [22.83 to NA] — Due to the limited number of events, the upper limit of the 95% CI for the median could not be derived.

3. Secondary Outcome: Locoregional Control (LRC) Time
Description: LRC time is defined as the time from randomization to the first occurrence of progression at the site of the primary tumor or the locoregional lymph nodes, either according to RECIST v1.1 or based on clinical assessment (radiological or clinical, as assessed by the Investigator). According to RECIST 1.1, progressive disease (PD) was defined as a 20% relative increase in the sum of diameters (SOD) of target lesions, taking as reference the nadir SOD and an absolute increase of >5 millimeter (mm) in the SOD, or the appearance of new lesions. Calculated via Kaplan Meier method.
Time Frame: From randomization to the first occurrence of progression at the site of the primary tumor or the locoregional lymph nodes or End Of Study (EOS) (188 weeks and 5 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 366
months | NA [0.0 to 37.0] — Due to the limited number of events, the median could not be derived. | NA [0.0 to 38.2] — Due to the limited number of events, the median could not be derived.

4. Secondary Outcome: Objective Response Rate (ORR) as Assessed by BIRC
Description: Objective response rate was defined as percentage of participants with either a confirmed complete response (CR) or partial response (PR). CR: Disappearance of all target and non-target lesions. PR: At least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum of their diameters, and no unequivocal progression of non-target lesions. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on the study, or unequivocal progression of non-target lesions, or appearance of any new lesion.
Time Frame: At 9 and 12 months post randomization
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 366
percentage of participants
  9 Months Post Randomization | 73.4 | 77.3
  12 Months Post Randomization | 73.6 | 77.9

5. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR defined as the number of participants with Complete Response by RECIST v1.1, as assessed by the BIRC. Complete response is defined as disappearance of all target and non-target lesions.
Time Frame: At 9 and 12 months post randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 366
Participants
  9 Months Post Randomization | 187 | 212
  12 Months Post Randomization | 194 | 222

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DoR) defined as the time from the first evidence of response (partial or complete, as assessed by the BIRC according to RECIST v1.1) to the first occurrence of progression (radiological or clinical, as assessed by the BIRC) or death from any cause. Kaplan Meier method was used for calculation.
Time Frame: Time from first evidence of response to the first occurrence of progression or death from any cause, assessed up to 24 months
Population: The ITT set included all randomized participants. Participants were analyzed according to the randomized treatment (assigned arm) assignment following the intention-to-treat principle. "Number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 269 | 287
months | NA [0.0 to 33.5] — Due to the limited number of events, the median could not be derived. | NA [0.0 to 33.7] — Due to the limited number of events, the median could not be derived.

7. Secondary Outcome: Number of Participants With Radical Salvage Surgery
Description: Number of Participants with Radical Salvage Surgery (excluding elective neck dissection without anatomopathological evidence of residual malignant cells) was reported.
Time Frame: At 9, 12, 24 and 36 months post randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 366
Participants
  Month 9 | 10 | 3
  Month 12 | 19 | 5
  Month 24 | 23 | 9
  Month 36 | 23 | 9

8. Secondary Outcome: Time to Subsequent Systemic Cancer Treatments
Description: Time to new subsequent systemic cancer treatment (in months) was derived as (date of event/censoring - randomization date +1) / 30.4375. Calculated via kaplan meier method.
Time Frame: Up to 188 weeks and 5 days post randomization
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 366
months | NA [NA to NA] — Median and 95% Confidence interval (CI) could not be calculated and estimated as there were insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated and estimated as there were insufficient number of participants with events.

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Adverse Events (AEs) of Special Interest
Description: An AE is any unfavorable/unintended sign (e.g., abnormal lab result), symptom or disease temporally linked to study drug, whether or not related. A serious AE leads to death, is life-threatening, causes significant/persistent disability, hospitalization, congenital anomaly, or is medically important. TEAEs include both serious and non-serious AEs after treatment. AESIs are events of clinical interest needing close monitoring. In this study, AESIs include: infusion reactions including hypersensitivity, immune-related AEs, aspartate aminotransferase/alanine transaminase increases, lipase/amylase elevation, acute renal failure, QTcF more than 30 milliseconds above baseline, and ≥Grade 2 inflammatory cutaneous AEs.
Time Frame: From signed informed consent to EOS (up to 188 weeks and 5 days)
Population: The safety analysis set (SAF set) included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT).
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
Participants
  TEAEs | 362 | 351
  Serious TEAEs | 194 | 129
  AESI | 357 | 342

10. Secondary Outcome: Number of Participants With Severity of Grade Greater or Equal to 3 TEAEs
Description: Severity of TEAEs were evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version. The grade are as follows: grade 1 : mild grade 2 : moderate grade 3 : severe or medically significant but not immediately life-threatening grade 4 : life threatening or disabling grade 5 : death related to AE.
Time Frame: From signed informed consent to EOS (up to 188 weeks and 5 days)
Population: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT).
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
Participants | 320 | 286

11. Secondary Outcome: Change From Baseline in Laboratory Parameters: Basophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Change from Baseline in Laboratory Parameters: Basophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets was reported.
Time Frame: At Baseline, Cycle 3 Day 1 (C3D1) (combination period), EOT (15 days after last study treatment administration) and baseline upto event free survival (EFS) follow up Month 18 after EOT (max on treatment change)
Population: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT). Here "overall number of participants analyzed signified" participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 363 | 352
10^9 cells per liter
  Basophils: Baseline | 0.052 (0.0343) | 0.054 (0.0367)
  Basophils: C3D1: number analyzed (Participants) | 283 | 288
  Basophils: C3D1 | -0.032 (0.0367) | -0.041 (0.0362)
  Basophils: EOT: number analyzed (Participants) | 280 | 287
  Basophils: EOT | -0.021 (0.0367) | -0.023 (0.0312)
  Basophil: Max on-treatment change: number analyzed (Participants) | 357 | 345
  Basophil: Max on-treatment change | -0.022 (0.0673) | -0.031 (0.0618)
  Leukocytes: Baseline | 8.175 (2.9656) | 8.105 (2.6725)
  Leukocytes: C3D1: number analyzed (Participants) | 288 | 290
  Leukocytes: C3D1 | -4.065 (3.1244) | -4.597 (2.9352)
  Leukocytes: EOT: number analyzed (Participants) | 282 | 287
  Leukocytes: EOT | -2.129 (3.2074) | -2.354 (2.4137)
  Leukocytes: Max on-treatment change: number analyzed (Participants) | 357 | 345
  Leukocytes: Max on-treatment change | -3.045 (7.5455) | -3.444 (6.7059)
  Lymphocytes: Baseline | 1.753 (0.5734) | 1.753 (0.6367)
  Lymphocytes: C3D1: number analyzed (Participants) | 283 | 288
  Lymphocytes: C3D1 | -1.168 (0.5804) | -1.251 (0.5742)
  Lymphocytes: EOT: number analyzed (Participants) | 280 | 287
  Lymphocytes: EOT | -0.884 (0.5485) | -0.901 (0.5536)
  Lymphocyte: Max on-treatment change: number analyzed (Participants) | 357 | 345
  Lymphocyte: Max on-treatment change | -1.382 (0.6359) | -1.356 (0.6150)
  Monocytes: Baseline | 0.518 (0.2156) | 0.506 (0.2072)
  Monocytes: C3D1: number analyzed (Participants) | 283 | 288
  Monocytes: C3D1 | -0.139 (0.2389) | -0.169 (0.2063)
  Monocytes: EOT: number analyzed (Participants) | 280 | 287
  Monocytes: EOT | -0.114 (0.1991) | -0.100 (0.1683)
  Monocyte: Max on-treatment change: number analyzed (Participants) | 357 | 345
  Monocyte: Max on-treatment change | -0.175 (0.4050) | -0.152 (0.3870)
  Neutrophils: Baseline | 5.669 (2.6589) | 5.610 (2.3663)
  Neutrophils: C3D1: number analyzed (Participants) | 283 | 288
  Neutrophils: C3D1 | -2.646 (2.8532) | -3.018 (2.6744)
  Neutrophils: EOT: number analyzed (Participants) | 280 | 287
  Neutrophils: EOT | -1.081 (2.9287) | -1.275 (2.2696)
  Neutrophils: Max on-treatment change: number analyzed (Participants) | 357 | 345
  Neutrophils: Max on-treatment change | -0.528 (7.2775) | -1.095 (6.3143)
  Platelets: Baseline: number analyzed (Participants) | 362 | 351
  Platelets: Baseline | 292.6 (104.86) | 287.7 (107.38)
  Platelets: C3D1: number analyzed (Participants) | 282 | 277
  Platelets: C3D1 | -48.2 (112.13) | -56.5 (109.52)
  Platelets: EOT: number analyzed (Participants) | 278 | 284
  Platelets: EOT | -24.8 (94.59) | -38.6 (87.16)
  Platelets: Max on-treatment change: number analyzed (Participants) | 356 | 344
  Platelets: Max on-treatment change | -63.2 (203.40) | -88.7 (171.61)

12. Secondary Outcome: Percent Change From Baseline in Laboratory Parameters: Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes, Neutrophils/Leukocytes
Description: Change from Baseline in Laboratory Parameters: Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes, Neutrophils/Leukocytes was reported.
Time Frame: At Cycle 3 Day 1 (C3D1) (combination period), EOT (15 days after last study treatment administration) and baseline upto event free survival (EFS) follow up Month 18 after EOT (max on treatment change)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 363 | 352
percent change
  C3D1: Basophils/Leukocytes: number analyzed (Participants) | 283 | 288
  C3D1: Basophils/Leukocytes | -0.21 (0.551) | -0.29 (0.527)
  EOT: Basophils/Leukocytes: number analyzed (Participants) | 280 | 287
  EOT: Basophils/Leukocytes | -0.14 (0.502) | -0.13 (0.483)
  Max on-treatment change: Basophils/Leukocytes: number analyzed (Participants) | 357 | 345
  Max on-treatment change: Basophils/Leukocytes | 0.03 (0.985) | 0.00 (1.032)
  C3D1: Eosinophils/Leukocytes: number analyzed (Participants) | 283 | 288
  C3D1: Eosinophils/Leukocytes | -0.04 (2.874) | -0.39 (2.147)
  EOT: Eosinophils/Leukocytes: number analyzed (Participants) | 280 | 287
  EOT: Eosinophils/Leukocytes | 0.60 (3.435) | 0.07 (1.878)
  Max on-treatment change: Eosinophils/Leukocytes: number analyzed (Participants) | 357 | 345
  Max on-treatment change: Eosinophils/Leukocytes | 1.32 (5.005) | 0.04 (3.308)
  C3D1: Lymphocytes/Leukocytes: number analyzed (Participants) | 283 | 288
  C3D1: Lymphocytes/Leukocytes | -6.89 (10.604) | -5.80 (10.086)
  EOT: Lymphocytes/Leukocytes: number analyzed (Participants) | 280 | 287
  EOT: Lymphocytes/Leukocytes | -6.85 (8.855) | -6.91 (7.850)
  Max on-treatment change: Lymphocytes/Leukocytes: number analyzed (Participants) | 357 | 345
  Max on-treatment change: Lymphocytes/Leukocytes | -11.39 (15.553) | -10.07 (15.985)
  C3D1: Monocytes/Leukocytes: number analyzed (Participants) | 283 | 288
  C3D1: Monocytes/Leukocytes | 3.65 (4.502) | 3.90 (3.840)
  EOT: Monocytes/Leukocytes: number analyzed (Participants) | 280 | 287
  EOT: Monocytes/Leukocytes | 0.64 (2.666) | 0.89 (2.454)
  Max on-treatment change: Monocytes/Leukocytes: number analyzed (Participants) | 357 | 345
  Max on-treatment change: Monocytes/Leukocytes | 5.87 (6.060) | 6.26 (5.631)
  C3D1: Neutrophils/Leukocytes: number analyzed (Participants) | 283 | 288
  C3D1: Neutrophils/Leukocytes | 2.67 (14.064) | 2.33 (12.467)
  EOT: Neutrophils/Leukocytes: number analyzed (Participants) | 280 | 287
  EOT: Neutrophils/Leukocytes | 5.75 (10.651) | 6.08 (9.086)
  Max on-treatment change: Neutrophils/Leukocytes: number analyzed (Participants) | 357 | 345
  Max on-treatment change: Neutrophils/Leukocytes | 6.80 (24.388) | 7.45 (21.764)

13. Secondary Outcome: Change From Baseline in Laboratory Parameters: Erythrocytes
Description: Change from Baseline in Laboratory Parameters: Erythrocytes was reported.
Time Frame: as for outcome 11
Population: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT). Here "overall number of participants analyzed" signified participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 363 | 352
10^12 cells per liter
  Baseline | 4.27 (0.507) | 4.37 (0.477)
  C3D1: number analyzed (Participants) | 288 | 290
  C3D1 | -0.81 (0.456) | -0.82 (0.433)
  EOT: number analyzed (Participants) | 282 | 287
  EOT | -0.70 (0.575) | -0.59 (0.464)
  Max on-treatment change: number analyzed (Participants) | 357 | 345
  Max on-treatment change | -1.14 (0.636) | -1.19 (0.605)

14. Secondary Outcome: Change From Baseline in Laboratory Parameters: Hemoglobin, Albumin, Protein
Description: Change from Baseline in Laboratory Parameters: Hemoglobin, Albumin, Protein was reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: grams per liters (g/L)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
grams per liters (g/L)
  Hemoglobin: Baseline: number analyzed (Participants) | 363 | 352
  Hemoglobin: Baseline | 132.9 (15.08) | 135.4 (14.34)
  Hemoglobin: C3D1: number analyzed (Participants) | 288 | 290
  Hemoglobin: C3D1 | -25.7 (14.24) | -25.2 (13.75)
  Hemoglobin: EOT: number analyzed (Participants) | 282 | 287
  Hemoglobin: EOT | -19.1 (17.73) | -14.4 (14.44)
  Hemoglobin: Max on-treatment change: number analyzed (Participants) | 357 | 345
  Hemoglobin: Max on-treatment change | -34.8 (19.83) | -35.8 (18.82)
  Albumin: Baseline: number analyzed (Participants) | 364 | 352
  Albumin: Baseline | 43.2 (3.95) | 43.6 (3.55)
  Albumin: C3D1: number analyzed (Participants) | 304 | 314
  Albumin: C3D1 | -4.0 (4.33) | -2.6 (3.61)
  Albumin: EOT: number analyzed (Participants) | 309 | 314
  Albumin: EOT | -1.1 (4.43) | 0.4 (4.02)
  Albumin: Max on-treatment change: number analyzed (Participants) | 351 | 343
  Albumin: Max on-treatment change | -4.8 (6.38) | -2.6 (5.90)
  Protein: Baseline: number analyzed (Participants) | 363 | 356
  Protein: Baseline | 70.1 (5.11) | 70.5 (4.78)
  Protein: C3D1: number analyzed (Participants) | 300 | 313
  Protein: C3D1 | -4.5 (5.73) | -4.3 (5.24)
  Protein: EOT: number analyzed (Participants) | 306 | 312
  Protein: EOT | -0.3 (6.10) | -0.7 (5.32)
  Protein: Max on-treatment change: number analyzed (Participants) | 350 | 343
  Protein: Max on-treatment change | -4.7 (9.12) | -5.0 (8.03)

15. Secondary Outcome: Change From Baseline in Laboratory Parameters: Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Aspartate Aminotransferase, Lipase
Description: Change from Baseline in Laboratory Parameters: Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Aspartate Aminotransferase, Lipase was reported.
Time Frame: as for outcome 11
Population: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT). Here "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
microgram per liter (mcg/L)
  Alanine Aminotransferase: Baseline: number analyzed (Participants) | 363 | 353
  Alanine Aminotransferase: Baseline | 18.9 (12.10) | 19.4 (12.66)
  Alanine Aminotransferase: C3D1: number analyzed (Participants) | 295 | 300
  Alanine Aminotransferase: C3D1 | 0.5 (16.77) | -4.6 (13.53)
  Alanine Aminotransferase: EOT: number analyzed (Participants) | 297 | 297
  Alanine Aminotransferase: EOT | -2.0 (18.25) | -3.4 (15.87)
  Alanine Aminotransferase: Max on-treatment change: number analyzed (Participants) | 356 | 346
  Alanine Aminotransferase: Max on-treatment change | 55.8 (70.73) | 26.5 (45.39)
  Alkaline Phosphatase: Baseline: number analyzed (Participants) | 363 | 356
  Alkaline Phosphatase: Baseline | 79.3 (24.48) | 78.0 (23.20)
  Alkaline Phosphatase: C3D1: number analyzed (Participants) | 301 | 312
  Alkaline Phosphatase: C3D1 | -0.8 (19.94) | -1.0 (21.89)
  Alkaline Phosphatase: EOT: number analyzed (Participants) | 305 | 311
  Alkaline Phosphatase: EOT | -2.2 (28.14) | -5.6 (18.79)
  Alkaline Phosphatase: Max on-treatment change: number analyzed (Participants) | 358 | 350
  Alkaline Phosphatase: Max on-treatment change | 12.7 (47.38) | 5.6 (49.27)
  Amylase: Baseline | 70.0 (42.81) | 67.8 (61.61)
  Amylase: C3D1: number analyzed (Participants) | 304 | 310
  Amylase: C3D1 | -14.0 (38.07) | -14.0 (32.85)
  Amylase: EOT: number analyzed (Participants) | 308 | 313
  Amylase: EOT | -13.5 (40.51) | -13.5 (33.79)
  Amylase: Max on-treatment change: number analyzed (Participants) | 359 | 350
  Amylase: Max on-treatment change | 125.8 (205.22) | 60.4 (119.29)
  Aspartate Aminotransferase: Baseline: number analyzed (Participants) | 363 | 356
  Aspartate Aminotransferase: Baseline | 19.8 (11.10) | 19.8 (8.31)
  Aspartate Aminotransferase: C3D1: number analyzed (Participants) | 302 | 311
  Aspartate Aminotransferase: C3D1 | -2.4 (12.30) | -3.5 (8.63)
  Aspartate Aminotransferase: EOT: number analyzed (Participants) | 304 | 312
  Aspartate Aminotransferase: EOT | 0.4 (19.01) | 0.9 (18.80)
  Aspartate Aminotransferase: Max on-treatment change: number analyzed (Participants) | 356 | 350
  Aspartate Aminotransferase: Max on-treatment change | 20.0 (37.35) | 9.7 (25.02)
  Lipase: Baseline | 35.4 (48.01) | 29.8 (19.37)
  Lipase: C3D1: number analyzed (Participants) | 305 | 309
  Lipase: C3D1 | -4.0 (39.69) | -4.0 (23.64)
  Lipase: EOT: number analyzed (Participants) | 308 | 314
  Lipase: EOT | -1.8 (47.38) | -1.0 (21.69)
  Lipase: Max on-treatment change: number analyzed (Participants) | 359 | 350
  Lipase: Max on-treatment change | 87.3 (196.87) | 25.0 (60.54)

16. Secondary Outcome: Change From Baseline in Laboratory Parameters: Bilirubin, Creatinine, Direct Bilirubin, Urate
Description: Change from Baseline in Laboratory Parameters: Bilirubin, Creatinine, Direct Bilirubin, Urate was reported.
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
micromole per liter (mcmol/L)
  Bilirubin: Baseline: number analyzed (Participants) | 364 | 355
  Bilirubin: Baseline | 7.4 (4.03) | 7.8 (4.06)
  Bilirubin: C3D1: number analyzed (Participants) | 304 | 312
  Bilirubin: C3D1 | -1.8 (3.74) | -1.5 (3.68)
  Bilirubin: EOT: number analyzed (Participants) | 309 | 314
  Bilirubin: EOT | -2.0 (3.85) | -1.3 (3.52)
  Bilirubin: Max on-treatment change: number analyzed (Participants) | 359 | 349
  Bilirubin: Max on-treatment change | 1.1 (7.49) | 0.1 (6.83)
  Creatinine: Baseline: number analyzed (Participants) | 363 | 356
  Creatinine: Baseline | 67.884 (15.1427) | 70.612 (15.3405)
  Creatinine: C3D1: number analyzed (Participants) | 301 | 312
  Creatinine: C3D1 | 11.771 (27.4012) | 11.740 (26.2545)
  Creatinine: EOT: number analyzed (Participants) | 306 | 313
  Creatinine: EOT | 17.660 (49.3934) | 16.243 (32.1216)
  Creatinine: Max on-treatment change: number analyzed (Participants) | 358 | 350
  Creatinine: Max on-treatment change | 292.808 (4199.9623) | 360.521 (5664.5213)
  Direct Bilirubin: Baseline: number analyzed (Participants) | 6 | 9
  Direct Bilirubin: Baseline | 4.8 (0.75) | 5.6 (1.33)
  Direct Bilirubin: C3D1: number analyzed (Participants) | 0 | 1
  Direct Bilirubin: C3D1 |  | 3.0 (NA) — Due to the presence of only a single data value for one participant, standard deviation could not be computed.
  Direct Bilirubin: EOT: number analyzed (Participants) | 0 | 2
  Direct Bilirubin: EOT |  | 0.0 (1.41)
  Direct Bilirubin: Max on-treatment change: number analyzed (Participants) | 2 | 8
  Direct Bilirubin: Max on-treatment change | 2.5 (2.12) | 1.0 (2.14)
  Urate: Baseline: number analyzed (Participants) | 363 | 356
  Urate: Baseline | 303.1 (79.62) | 305.9 (82.79)
  Urate: C3D1: number analyzed (Participants) | 301 | 313
  Urate: C3D1 | -25.4 (90.93) | -21.5 (91.07)
  Urate: EOT: number analyzed (Participants) | 306 | 313
  Urate: EOT | 25.9 (85.01) | 33.1 (80.07)
  Urate: Max on-treatment change: number analyzed (Participants) | 350 | 343
  Urate: Max on-treatment change | 1.2 (140.44) | 12.7 (137.74)

17. Secondary Outcome: Change From Baseline in Laboratory Parameters: C Reactive Protein
Description: Change from Baseline in Laboratory Parameters: C Reactive Protein was reported.
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
milligrams per liter (mg/L)
  Baseline | 15.80 (24.655) | 13.78 (21.780)
  C3D1: number analyzed (Participants) | 304 | 307
  C3D1 | 25.30 (50.259) | 11.66 (36.791)
  EOT: number analyzed (Participants) | 306 | 314
  EOT | 1.26 (31.784) | 1.22 (27.720)
  Max on-treatment change: number analyzed (Participants) | 351 | 343
  Max on-treatment change | 43.91 (66.024) | 27.90 (56.262)

18. Secondary Outcome: Change From Baseline in Laboratory Parameters: Calcium, Magnesium, Potassium, Sodium, Urea
Description: Change from Baseline in Laboratory Parameters: Calcium, Magnesium, Potassium, Sodium, Urea was reported.
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
millimoles per liter (mmol/L)
  Calcium: Baseline | 2.4065 (0.14050) | 2.4043 (0.11777)
  Calcium: C3D1: number analyzed (Participants) | 304 | 314
  Calcium: C3D1 | -0.1054 (0.16830) | -0.0574 (0.12989)
  Calcium: EOT: number analyzed (Participants) | 309 | 314
  Calcium: EOT | 0.0006 (0.15586) | 0.0136 (0.12258)
  Calcium: Max on-treatment change: number analyzed (Participants) | 351 | 346
  Calcium: Max on-treatment change | -0.1182 (0.64226) | -0.0575 (0.63941)
  Magnesium: Baseline: number analyzed (Participants) | 363 | 356
  Magnesium: Baseline | 0.8731 (0.08816) | 0.8718 (0.08800)
  Magnesium: C3D1: number analyzed (Participants) | 301 | 313
  Magnesium: C3D1 | -0.0871 (0.11743) | -0.0719 (0.11889)
  Magnesium: EOT: number analyzed (Participants) | 306 | 313
  Magnesium: EOT | -0.0588 (0.10612) | -0.0372 (0.08725)
  Magnesium: Max on-treatment change: number analyzed (Participants) | 350 | 345
  Magnesium: Max on-treatment change | -0.1231 (0.21711) | -0.0860 (0.21948)
  Potassium: Baseline: number analyzed (Participants) | 363 | 356
  Potassium: Baseline | 4.4270 (0.41610) | 4.4534 (0.44584)
  Potassium: C3D1: number analyzed (Participants) | 301 | 309
  Potassium: C3D1 | -0.1226 (0.60007) | -0.0877 (0.58424)
  Potassium: EOT: number analyzed (Participants) | 302 | 311
  Potassium: EOT | -0.0374 (0.52898) | 0.0170 (0.58221)
  Potassium: Max on-treatment change: number analyzed (Participants) | 356 | 350
  Potassium: Max on-treatment change | -0.2845 (1.13356) | -0.2551 (1.14282)
  Sodium: Baseline: number analyzed (Participants) | 363 | 356
  Sodium: Baseline | 139.3333 (2.72935) | 139.1798 (3.19705)
  Sodium: C3D1: number analyzed (Participants) | 302 | 313
  Sodium: C3D1 | -2.0828 (3.96368) | -1.5527 (3.73110)
  Sodium: EOT: number analyzed (Participants) | 306 | 313
  Sodium: EOT | -0.9510 (3.53728) | -0.9521 (3.71944)
  Sodium: Max on-treatment change: number analyzed (Participants) | 358 | 350
  Sodium: Max on-treatment change | -4.7482 (9.86512) | -4.6627 (14.14911)
  Urea: Baseline: number analyzed (Participants) | 363 | 356
  Urea: Baseline | 5.22 (1.885) | 5.23 (2.068)
  Urea: C3D1: number analyzed (Participants) | 302 | 312
  Urea: C3D1 | 1.89 (3.302) | 1.87 (3.961)
  Urea: EOT: number analyzed (Participants) | 306 | 313
  Urea: EOT | 1.73 (3.266) | 1.40 (2.922)
  Urea: Max on-treatment change: number analyzed (Participants) | 358 | 350
  Urea: Max on-treatment change | 8.51 (7.226) | 6.18 (6.110)

19. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate
Description: Change from baseline in biochemistry parameter eGFR was reported. The Glomerular Filtration Rate was measured as milliliter per minute per 1.73 square meter (mL/min/1.73m^2).
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/min/1.73m*2
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 361 | 356
mL/min/1.73m*2
  Baseline | 96.956 (14.2212) | 95.244 (14.1290)
  C3D1: number analyzed (Participants) | 299 | 312
  C3D1 | -8.799 (19.0295) | -9.205 (18.5178)
  EOT: number analyzed (Participants) | 304 | 313
  EOT | -11.385 (20.6015) | -12.594 (18.0053)
  Max on-treatment change: number analyzed (Participants) | 348 | 346
  Max on-treatment change | -19.439 (27.3672) | -19.528 (25.7099)

20. Secondary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (PTT)/ Standard and Prothrombin Time
Description: Change from Baseline in coagulation parameter activated PTT/standard and prothrombin Time was reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: seconds (Sec)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 349 | 344
seconds (Sec)
  Activated PTT/Standard: Baseline: number analyzed (Participants) | 347 | 340
  Activated PTT/Standard: Baseline | 26.15 (2.349) | 26.25 (2.540)
  Activated PTT/Standard: C3D1: number analyzed (Participants) | 269 | 273
  Activated PTT/Standard: C3D1 | -0.80 (3.132) | -0.91 (2.324)
  Activated PTT/Standard: EOT: number analyzed (Participants) | 260 | 268
  Activated PTT/Standard: EOT | -0.29 (2.812) | -0.09 (2.419)
  Activated PTT/Standard: Max on-treatment change: number analyzed (Participants) | 331 | 322
  Activated PTT/Standard: Max on-treatment change | -1.01 (4.165) | -0.87 (3.509)
  Prothrombin Time: Baseline | 10.50 (0.730) | 10.73 (1.696)
  Prothrombin Time: C3D1: number analyzed (Participants) | 274 | 284
  Prothrombin Time: C3D1 | 0.11 (1.730) | -0.17 (1.543)
  Prothrombin Time: EOT: number analyzed (Participants) | 266 | 283
  Prothrombin Time: EOT | 0.17 (1.757) | -0.04 (1.697)
  Prothrombin Time: Max on-treatment change: number analyzed (Participants) | 334 | 329
  Prothrombin Time: Max on-treatment change | 0.35 (2.364) | -0.01 (1.838)

21. Secondary Outcome: Change From Baseline in Fibrinogen
Description: Change from Baseline in coagulation parameter fibrinogen was reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dl)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 348 | 343
milligrams per deciliter (mg/dl)
  Baseline | 486.9 (140.35) | 467.7 (119.14)
  C3D1: number analyzed (Participants) | 273 | 282
  C3D1 | 121.3 (164.05) | 109.8 (157.03)
  EOT: number analyzed (Participants) | 265 | 283
  EOT | 17.8 (150.78) | 1.0 (138.69)
  Max on-treatment change: number analyzed (Participants) | 333 | 328
  Max on-treatment change | 112.6 (212.46) | 122.4 (207.11)

22. Secondary Outcome: Change From Baseline in Prothrombin International Normalized Ratio
Description: Change from baseline in coagulation parameters prothrombin international normalized ratio was reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 349 | 344
ratio
  Baseline | 0.96 (0.090) | 0.99 (0.188)
  C3D1: number analyzed (Participants) | 274 | 284
  C3D1 | 0.01 (0.195) | -0.02 (0.175)
  EOT: number analyzed (Participants) | 266 | 283
  EOT | 0.02 (0.197) | 0.00 (0.195)
  Max on-treatment change: number analyzed (Participants) | 334 | 329
  Max on-treatment change | 0.04 (0.265) | 0.00 (0.212)

23. Secondary Outcome: Change From Baseline in Vital Signs: Systolic Blood Pressure, Diastolic Blood Pressure
Description: Change from Baseline in Vital Signs: Systolic Blood Pressure, Diastolic Blood Pressure was reported.
Time Frame: At Baseline, Cycle 3 Day 1 (C3D1) (combination period), EOT (15 days after last study treatment administration) and baseline upto event free survival (EFS) follow up Month 18 after EOT (max on treatment increase & decrease)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
millimeters of mercury (mmHg)
  Systolic Blood Pressure: Baseline | 128.0 (18.08) | 128.2 (16.96)
  Systolic Blood Pressure: C3D1: number analyzed (Participants) | 320 | 326
  Systolic Blood Pressure: C3D1 | -10.1 (19.36) | -7.9 (17.53)
  Systolic Blood Pressure: EOT: number analyzed (Participants) | 320 | 323
  Systolic Blood Pressure: EOT | -5.8 (20.47) | -3.4 (20.03)
  Systolic BP: Max on-treatment increase: number analyzed (Participants) | 249 | 274
  Systolic BP: Max on-treatment increase | 15.6 (12.89) | 16.5 (12.43)
  Systolic BP: Max on-treatment decrease: number analyzed (Participants) | 328 | 323
  Systolic BP: Max on-treatment decrease | -24.7 (15.85) | -21.9 (14.48)
  Diastolic Blood Pressure: Baseline | 77.4 (10.60) | 77.5 (9.75)
  Diastolic Blood Pressure: C3D1: number analyzed (Participants) | 320 | 326
  Diastolic Blood Pressure: C3D1 | -5.6 (12.04) | -4.0 (10.65)
  Diastolic Blood Pressure: EOT: number analyzed (Participants) | 320 | 323
  Diastolic Blood Pressure: EOT | -1.8 (12.02) | -1.2 (11.55)
  Diastolic BP: Max on-treatment increase: number analyzed (Participants) | 241 | 250
  Diastolic BP: Max on-treatment increase | 11.1 (7.54) | 11.2 (8.09)
  Diastolic BP: Max on-treatment decrease: number analyzed (Participants) | 323 | 319
  Diastolic BP: Max on-treatment decrease | -15.2 (9.43) | -13.2 (8.42)

24. Secondary Outcome: Change From Baseline in Vital Signs: Heart Rate
Description: Change from Baseline in Vital Signs: Heart Rate was reported.
Time Frame: as for outcome 23
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
beats/minute
  Heart Rate: Baseline | 77.6 (12.35) | 76.1 (12.60)
  Heart Rate: C3D1: number analyzed (Participants) | 320 | 326
  Heart Rate: C3D1 | 5.2 (13.71) | 3.4 (13.92)
  Heart Rate: EOT: number analyzed (Participants) | 318 | 323
  Heart Rate: EOT | 2.8 (14.33) | 2.2 (13.51)
  Heart Rate: Max on-treatment increase: number analyzed (Participants) | 316 | 304
  Heart Rate: Max on-treatment increase | 17.8 (12.30) | 16.7 (10.97)
  Heart Rate: Max on-treatment decrease: number analyzed (Participants) | 274 | 280
  Heart Rate: Max on-treatment decrease | -11.7 (9.00) | -12.2 (9.13)

25. Secondary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: Change from Baseline in Vital Signs: Respiratory Rate was reported.
Time Frame: as for outcome 23
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 359 | 355
breaths/minute
  Respiratory Rate: Baseline | 16.8 (2.38) | 16.7 (2.98)
  Respiratory Rate: C3D1: number analyzed (Participants) | 304 | 319
  Respiratory Rate: C3D1 | -0.1 (2.65) | 0.0 (2.76)
  Respiratory Rate: EOT: number analyzed (Participants) | 308 | 317
  Respiratory Rate: EOT | -0.1 (2.83) | -0.1 (3.01)
  Respiratory Rate: Max on-treatment increase: number analyzed (Participants) | 208 | 216
  Respiratory Rate: Max on-treatment increase | 3.2 (2.66) | 2.7 (2.13)
  Respiratory Rate: Max on-treatment decrease: number analyzed (Participants) | 208 | 216
  Respiratory Rate: Max on-treatment decrease | -3.1 (2.52) | -2.7 (2.88)

26. Secondary Outcome: Change From Baseline in Vital Signs: Body Temperature
Description: Change from Baseline in Vital Signs: Body Temperature was reported.
Time Frame: At Baseline, Cycle 3 Day 1 (C3D1) (combination period), EOT (15 days after last study treatment administration) and baseline upto event free survival (EFS) follow up Month 18 after EOT (max on treatment increase)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 355
degree Celsius
  Baseline | 36.44 (0.443) | 36.41 (0.432)
  C3D1: number analyzed (Participants) | 318 | 325
  C3D1 | 0.10 (36.49) | 0.07 (0.476)
  EOT: number analyzed (Participants) | 317 | 320
  EOT | 0.00 (0.463) | 0.00 (0.453)
  Max on-treatment increase: number analyzed (Participants) | 292 | 295
  Max on-treatment increase | 0.57 (0.445) | 0.51 (0.413)

27. Secondary Outcome: Change From Baseline in Vital Signs: Body Weight
Description: Change from Baseline in Vital Signs: Body Weight was reported.
Time Frame: At Baseline, C3D1 (combination period), EOT (15 days after last study treatment administration) and baseline upto event free survival (EFS) follow up Month 18 after EOT (max on treatment increase & decrease)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
kilograms (kg)
  Baseline | 69.552 (16.8493) | 70.261 (15.2793)
  C3D1: number analyzed (Participants) | 321 | 327
  C3D1 | -4.762 (3.9129) | -4.331 (3.6001)
  EOT: number analyzed (Participants) | 319 | 328
  EOT | -6.282 (6.1160) | -4.819 (5.9718)
  Max on-treatment increase: number analyzed (Participants) | 86 | 104
  Max on-treatment increase | 2.497 (2.1157) | 2.549 (2.7503)
  Max on-treatment decrease: number analyzed (Participants) | 340 | 331
  Max on-treatment decrease | -8.182 (5.1605) | -7.379 (4.8001)

28. Secondary Outcome: Change From Baseline in ECG Parameters
Description: The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. The parameters included Respiratory Rate (RR), Pulse Rate (PR), QRS, QT and QTcF calculated by the Bazett formula.
Time Frame: At Baseline, and upto event free survival (EFS) follow up Month 18 after EOT (max on treatment increase)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
millisecond
  PR Interval: Baseline: number analyzed (Participants) | 361 | 353
  PR Interval: Baseline | 154.6 (28.05) | 159.2 (29.85)
  PR Interval: Max on-treatment increase: number analyzed (Participants) | 273 | 247
  PR Interval: Max on-treatment increase | 15.2 (16.48) | 15.8 (19.90)
  QRS Duration: Baseline: number analyzed (Participants) | 364 | 355
  QRS Duration: Baseline | 90.4 (14.78) | 91.9 (14.48)
  QRS Duration: Max on-treatment increase: number analyzed (Participants) | 267 | 268
  QRS Duration: Max on-treatment increase | 9.8 (9.87) | 9.8 (21.97)
  QT Interval: Baseline | 381.9 (30.29) | 385.7 (33.47)
  QT Interval: Max on-treatment increase: number analyzed (Participants) | 307 | 278
  QT Interval: Max on-treatment increase | 33.3 (26.91) | 26.9 (21.78)
  RR Interval: Baseline: number analyzed (Participants) | 359 | 349
  RR Interval: Baseline | 824.5 (163.43) | 858.0 (153.30)
  RR Interval: Max on-treatment increase: number analyzed (Participants) | 291 | 266
  RR Interval: Max on-treatment increase | 139.5 (125.19) | 117.2 (87.11)
  QTcF Interval: Baseline | 406.3 (22.78) | 406.6 (25.06)
  QTcF Interval: Max on-treatment increase: number analyzed (Participants) | 305 | 279
  QTcF Interval: Max on-treatment increase | 24.9 (21.27) | 19.7 (19.17)

29. Secondary Outcome: Treatment Duration
Description: Treatment duration is calculated by study treatment component as (last dose date minus first dose date plus x)/7, where x=8 for xevinapant/matched placebo, x=21 for cisplatin/carboplatin, x=3 for IMRT.
Time Frame: Up to end of study (up to 188weeks and 5 days)
Population: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT). Here "number analyzed" signifies participants who were evaluable for each specific category.
Measure: Median (Full Range); unit: weeks
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
weeks
  Xevinapant/matched placebo | 18.00 [10.71 to 18.14] | 18.00 [18.00 to 18.29]
  Cisplatin: number analyzed (Participants) | 360 | 351
  Cisplatin | 8.86 [6.00 to 9.00] | 9.00 [6.00 to 9.00]
  Carboplatin: number analyzed (Participants) | 55 | 60
  Carboplatin | 3.00 [3.00 to 6.00] | 3.00 [3.00 to 6.00]
  IMRT: number analyzed (Participants) | 364 | 355
  IMRT | 7.43 [7.21 to 7.86] | 7.43 [7.29 to 7.71]

30. Secondary Outcome: Number of Participants Who Completed Cycle 1, 2, 3, 4, 5 and 6
Description: Number of participants who completed cycle 1, 2, 3, 4, 5 or 6 of xevinapant/matched placebo were reported.
Time Frame: Cycle 1, 2, 3, 4, 5 and 6 (each cycle is of 3 weeks)
Population: as for outcome 10
Measure: Number; unit: count of participants
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
count of participants
  Cycle 1 | 363 | 355
  Cycle 2 | 325 | 335
  Cycle 3 | 290 | 314
  Cycle 4 | 266 | 210
  Cycle 5 | 263 | 307
  Cycle 6 | 246 | 297

31. Secondary Outcome: Total Cumulative Dose of Xevinapant/ Matched Placebo
Description: Total cumulative dose of Xevinapant/ Matched Placebo was reported in form of mean and standard deviation.
Time Frame: Up to end of treatment (Day 134)
Population: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT). Here "overall number of participants analyzed signified" participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 355
milligrams (mg) | 12383.6 (5375.66) | 14417.0 (4288.55)

32. Secondary Outcome: Total Cumulative Dose of Cisplatin
Description: Total cumulative dose of cisplatin was reported.
Time Frame: Up to end of treatment (Day 134)
Population: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT). Here" overall number of participants analyzed signified" participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per square meter (mg/m^2)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 360 | 351
milligrams per square meter (mg/m^2) | 223.3 (76.26) | 236.3 (73.14)

33. Secondary Outcome: Total Cumulative Dose of Carboplatin
Description: Total cumulative dose of carboplatin was reported as mean and standard deviation.
Time Frame: Up to end of treatment (Day 134)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mg*min/mL
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 54 | 60
mg*min/mL | 6.9 (2.37) | 6.6 (2.26)

34. Secondary Outcome: Total Cumulative Dose of Intensity-Modulated Radiation Therapy (IMRT)
Description: Total cumulative dose of IMRT were reported in form of mean and standard deviation.
Time Frame: Up to end of treatment (Day 134)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Gray (Gy)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 355
Gray (Gy) | 66.4 (12.32) | 67.9 (9.74)

35. Secondary Outcome: Overall Dose Intensity of Xevinapant/Matched Placebo
Description: Overall dose intensity of Xevinapant/ matched placebo is calculated as the mean of the dose intensities of the individual cycles.
Time Frame: Cycle 1, 2, 3, 4 5, 6 (each cycle is of 3 weeks) or End of Treatment (Day 134)
Population: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT).Here "overall number of participants analyzed signified" participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per day (mg/day)
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 355
milligrams per day (mg/day) | 122.72 (18.274) | 126.56 (16.495)

36. Secondary Outcome: Overall Dose Intensity of Cisplatin
Description: Overall dose intensity of Cisplatin is calculated as the mean of the dose intensities of the individual cycles. This was reported with the unit of measure milligrams per meter square per week (mg/m2/week).
Time Frame: Cycle 1, 2, 3, 4 5, 6 (each cycle is of 3 weeks) or End of Treatment (Day 134)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mg/m2/week
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 360 | 351
mg/m2/week | 32.33 (3.053) | 32.55 (2.301)

37. Secondary Outcome: Overall Dose Intensity of Carboplatin
Description: Overall dose intensity of Carboplatin is calculated as the mean of the dose intensities of the individual cycles. This was reported with unit of measure Milligrams per minute per milliliter per week (mg min/mL/week).
Time Frame: Cycle 1, 2, 3, 4 5, 6 (each cycle is of 3 weeks) or End of Treatment (Day 134)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mg min/mL/week
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 54 | 60
mg min/mL/week | 1.59 (0.136) | 1.60 (0.123)

38. Secondary Outcome: Relative Dose Intensity
Description: Relative dose intensity (RDI) represents the percentage of the amount of a drug actually delivered [actual dose intensity (DI)] to the amount planned (planned DI). The purpose of calculating RDI is to evaluate whether the planned DI of an anti-cancer treatment was actually achieved which may suggest the feasibility of planned treatment regimen.
Time Frame: Up to 50 months
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percentage (%) of dose intensity
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 363 | 355
percentage (%) of dose intensity
  Xevinapant/matched placebo | 92.04 (13.706) | 94.92 (12.372)
  Cisplatin: number analyzed (Participants) | 360 | 351
  Cisplatin | 96.98 (9.159) | 97.65 (6.904)
  Carboplatin: number analyzed (Participants) | 54 | 60
  Carboplatin | 95.19 (8.182) | 96.17 (7.386)

39. Secondary Outcome: Number of Participants With Treatment Interruption, Treatment Reduction and Treatment Discontinuation for Xevinapant/ Matched Placebo
Description: Number of participants with Treatment Interruption, Treatment Reduction and Treatment Discontinuation was reported.
Time Frame: Up to end of treatment (Day 134)
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 356
Participants
  Treatment Interruption of xevinapant/ matched placebo | 206 | 147
  Treatment Reduction of xevinapant/ matched placebo | 34 | 17
  Treatment Discontinuation of xevinapant/ matched placebo | 71 | 30

40. Primary Outcome: Event-Free Survival (EFS) as Assessed by Blinded Independent Review Committee (BIRC)
Description: Event-Free Survival (EFS) as assessed by BIRC is the time from randomization to the first of: (1) Death from any cause; (2) Progression: either radiological (per RECIST v1.1) or clinical (with/without radiologic proof, assessed endoscopically); (3) Primary treatment failure prior to complete response (CR): requirement for radical salvage surgery at primary tumor site with viable tumor confirmed histologically, even without RECIST progression; (4) Relapse after CR (locoregional): including radical salvage surgery or elective neck dissection/biopsy more than equal to (>=) 22 weeks post-randomization showing viable tumor cells regardless of radiologic status; (5) Second cancers, unless histology excludes squamous origin. Calculated via Kaplan Meier method.
Time Frame: From randomization to the earliest between any EFS event or End of Study (EOS) (up to 188 weeks and 5 days)
Population: The Intention To Treat (ITT) set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
Number analyzed (Participants) | 364 | 366
months | 19.4 [14.46 to NA] — Due to the limited number of events, the upper limit of the 95% CI for the median could not be derived. | 33.1 [20.99 to NA] — Due to the limited number of events, the upper limit of the 95% CI for the median could not be derived.

ADVERSE EVENTS:
Time Frame: All AEs and All-Cause Mortality were be collected from the time of Informed Consent Form signature until the End Of Treatment (EOT) visit (Day 134) . From the EOT visit until the End Of Study visit (Up to 44 months), only All-Cause Mortality, SAEs and late onset Adverse Events of Special Interest were collected
Description: The SAF set included all participants who received any dose of any of the study intervention (xevinapant/matched placebo, cisplatin/carboplatin, IMRT) and All-Cause Mortality was assessed in all enrolled participants.
Arm/Group | Sequence 1: Debio 1143 + CRT | Sequence 2: Placebo + CRT
All-Cause Mortality (participants affected / at risk) | 111/364 | 93/366
Serious Adverse Events (participants affected / at risk) | 194/364 | 129/356
Other Adverse Events (participants affected / at risk) | 360/364 | 350/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1: Debio 1143 + CRT (N=364) | Sequence 2: Placebo + CRT (N=356)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 7 (7)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 8 (8)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ototoxicity (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Central hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 9 (9) | 21 (21)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (9) | 5 (5)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 5 (5)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 15 (16)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 6 (6)
Asthenia (General disorders) | 2 (2) | 5 (5)
Death (General disorders) | 2 (2) | 2 (2)
Disease progression (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 8 (8)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 5 (7)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Epiglottic abscess (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (14) | 23 (24)
Pneumonia aspiration (Infections and infestations) | 4 (4) | 8 (9)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 3 (3) | 8 (8)
Stoma site infection (Infections and infestations) | 0 (0) | 5 (5)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site discharge (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 5 (5) | 12 (12)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 4 (4)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 4 (4)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 7 (8)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 2 (2)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Diplegia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 19 (20) | 25 (31)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 6 (7) | 10 (11)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vein thrombus extension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1: Debio 1143 + CRT (N=364) | Sequence 2: Placebo + CRT (N=356)
Anaemia (Blood and lymphatic system disorders) | 180 (212) | 199 (244)
Leukopenia (Blood and lymphatic system disorders) | 44 (69) | 57 (79)
Lymphopenia (Blood and lymphatic system disorders) | 42 (46) | 39 (48)
Neutropenia (Blood and lymphatic system disorders) | 100 (136) | 110 (141)
Thrombocytopenia (Blood and lymphatic system disorders) | 45 (61) | 63 (79)
Deafness (Ear and labyrinth disorders) | 18 (18) | 19 (19)
Hypoacusis (Ear and labyrinth disorders) | 30 (33) | 21 (21)
Tinnitus (Ear and labyrinth disorders) | 65 (70) | 59 (67)
Constipation (Gastrointestinal disorders) | 125 (146) | 126 (144)
Diarrhoea (Gastrointestinal disorders) | 46 (51) | 40 (44)
Dry mouth (Gastrointestinal disorders) | 124 (131) | 138 (143)
Dysphagia (Gastrointestinal disorders) | 97 (103) | 138 (154)
Nausea (Gastrointestinal disorders) | 162 (238) | 144 (188)
Odynophagia (Gastrointestinal disorders) | 77 (84) | 66 (69)
Salivary hypersecretion (Gastrointestinal disorders) | 12 (13) | 20 (20)
Stomatitis (Gastrointestinal disorders) | 160 (173) | 193 (224)
Vomiting (Gastrointestinal disorders) | 84 (112) | 66 (85)
Asthenia (General disorders) | 68 (88) | 98 (108)
Fatigue (General disorders) | 66 (75) | 58 (71)
Pyrexia (General disorders) | 35 (42) | 58 (72)
COVID-19 (Infections and infestations) | 22 (22) | 27 (27)
Oral candidiasis (Infections and infestations) | 20 (26) | 18 (19)
Radiation mucositis (Injury, poisoning and procedural complications) | 23 (23) | 20 (20)
Radiation skin injury (Injury, poisoning and procedural complications) | 160 (166) | 165 (175)
Alanine aminotransferase increased (Investigations) | 40 (54) | 78 (115)
Amylase increased (Investigations) | 44 (50) | 84 (110)
Aspartate aminotransferase increased (Investigations) | 30 (43) | 47 (56)
Blood creatinine increased (Investigations) | 81 (106) | 87 (119)
Blood urea increased (Investigations) | 17 (28) | 20 (27)
C-reactive protein increased (Investigations) | 17 (21) | 24 (26)
Electrocardiogram QT prolonged (Investigations) | 14 (14) | 26 (29)
Gamma-glutamyltransferase increased (Investigations) | 19 (22) | 23 (26)
Lipase increased (Investigations) | 23 (32) | 56 (76)
Lymphocyte count decreased (Investigations) | 30 (39) | 45 (63)
Neutrophil count decreased (Investigations) | 76 (122) | 78 (118)
Platelet count decreased (Investigations) | 46 (71) | 57 (82)
Weight decreased (Investigations) | 157 (171) | 187 (201)
White blood cell count decreased (Investigations) | 65 (127) | 63 (113)
Decreased appetite (Metabolism and nutrition disorders) | 97 (115) | 65 (76)
Dehydration (Metabolism and nutrition disorders) | 17 (22) | 19 (20)
Hyperkalaemia (Metabolism and nutrition disorders) | 17 (21) | 25 (34)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 22 (30) | 31 (40)
Hypocalcaemia (Metabolism and nutrition disorders) | 12 (14) | 26 (36)
Hypokalaemia (Metabolism and nutrition disorders) | 63 (83) | 71 (103)
Hypomagnesaemia (Metabolism and nutrition disorders) | 43 (52) | 54 (64)
Hyponatraemia (Metabolism and nutrition disorders) | 42 (49) | 64 (97)
Neck pain (Musculoskeletal and connective tissue disorders) | 21 (21) | 20 (23)
Dizziness (Nervous system disorders) | 18 (19) | 20 (22)
Dysgeusia (Nervous system disorders) | 111 (117) | 106 (109)
Headache (Nervous system disorders) | 22 (24) | 23 (24)
Insomnia (Psychiatric disorders) | 26 (27) | 37 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (48) | 36 (38)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 42 (45) | 36 (38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 19 (22)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 28 (33) | 21 (24)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 62 (65) | 56 (60)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 21 (23)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 23 (23)
Dermatitis (Skin and subcutaneous tissue disorders) | 54 (58) | 57 (60)
Rash (Skin and subcutaneous tissue disorders) | 13 (15) | 40 (49)
Hypertension (Vascular disorders) | 20 (26) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT04459715/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04459715/SAP_001.pdf